CLINICAL TRIAL: NCT03762395
Title: Anti Inflammatory Lipid Mediators in Asthma: A Double Blind Placebo Control Cross Over, Proof of Concept Study of CXA-10 to Reduce Bronchial Hyperresponsiveness in Obese Asthmatics; Lipid Anti-Inflammatory Mediators in Asthma to Reduce Hyperresponsiveness in Obese Asthmatics
Brief Title: Anti Inflammatory Lipid Mediators in Asthma Lipid Anti-Inflammtory Mediators in Asthma
Acronym: ALMA; LIMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0510; 21-3959; 5R01HL132550-03 (NIH); 1R61HL157069-01A1 (NIH)
Record Dates: First submitted 2018-08-01; First posted 2018-12-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — CXA-10

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CXA-10 (Experimental): Administered orally, continuously, and daily for at least 6 weeks. Dispensed at Visit 1. Washout period of at least 4 weeks and then enter crossover phase of an additional 6 weeks. Drug will be dispensed at Visit 4.
  Interventions: Drug: CXA-10
- Matching Placebo (Placebo Comparator): Administered orally, daily, and continuously for at least 6 weeks. Dispensed at Visit 1. Washout period of at least 4 weeks and then enter crossover phase of an additional 6 weeks. Placebo will be dispensed at Visit 4.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CXA-10 — 6 weeks of treatment with 150 mg/day of orally administered CXA-10
  Other Names: 10-nitro-9(E)-octadec-9-enoic acid
  Arms: CXA-10
Drug: Matching Placebo — 6 weeks of treatment with orally administered matching placebo (to 150 mg/day of CXA-10)
  Arms: Matching Placebo

SUMMARY:
The main purpose of this Phase 2 double blind, placebo controlled crossover clinical study is to demonstrate the efficacy and safety of CXA-10 in obese adult asthmatics. Obesity induces a chronic systemic inflammatory state characterized by impaired adipokine signaling, pro-inflammatory cytokine responses, inflammatory cell activation and enhanced generation of oxidative inflammatory mediators. This impacts the lung, increasing the severity of asthma and its exacerbations. This research will evaluate how a synthetic nitro-fatty acid (CXA-10, 10-nitro-octadec-9-enoic acid) suppresses the systemic and airway inflammation that contributes to the obese asthmatic phenotype. Current data support the pleiotropic signaling actions of CXA-10 to induce adaptive signaling actions that beneficially modulate adipokine and cytokine expression and inhibit systemic and pulmonary inflammation. The investigators hypothesize that CXA-10 induced signaling responses will alleviate obesity-related airway hyperreactivity in obese adult asthmatics.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate completion of informed consent process with written documentation. Male and female patients, 18 to 65 years old. Female subjects should be either post-menopausal or surgically sterile, or, if child-bearing potential (WOCP) should agree to use an acceptable method of contraception, for the duration of the study, with a negative pregnancy test prior to entering the study.
2. BMI >/= 30
3. Diagnosis of asthma: based on previous physician diagnosis for > 6 months, and baseline pre-bronchodilator (BD) FEV1 between 50 and 95% predicted with either a 12% or greater bronchodilator response to 4 puffs of albuterol or PC20 methacholine (16 mg) if <12% change post BD
4. Regular treatment with inhaled corticosteroids (ICS) (up to 1000 mcg/day fluticasone/equivalent), long acting beta agonists (LABA), and/or long-acting muscarinic antagonists (LAMA), which can be combination medication for at least 3 months; on a stable dose for the 4 weeks prior to Visit 0

Exclusion Criteria:

1. Respiratory tract infection within the last 4 weeks
2. Oral or systemic corticosteroid burst within the last 4 weeks
3. Asthma-related hospitalization within the last 6 weeks
4. Three or more asthma exacerbations requiring treatment with systemic corticosteroids in the past year consistent with severe asthma
5. Asthma-related ER visit within the previous 4 weeks
6. Current smoking or have former smokers that quit within the previous 1 year, or 10 pack years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Methacholine challenge dose per spirometry | Through study completion, up to 18 weeks
  To determine CXA-10 efficacy, reduction of bronchial hyperresponsiveness determined by performing spirometry to see if there's a change in methacholine dose
Changes in pre-bronchodilator FEV1 per spirometry | Through study completion, up to 18 weeks
  To determine the efficacy of CXA-10 by improving FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver- Anschutz Medical Campus
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No